CLINICAL TRIAL: NCT04286451
Title: Effect of Sleep Restriction on Adipose Tissue and Skeletal Muscle Insulin Sensitivity
Acronym: SLEEP-IN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Prachi Singh, Associate Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: PBRC 2020-007
Record Dates: First submitted 2020-01-13; First posted 2020-02-27 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Sleep Disturbance; Postmenopausal Symptoms; Insulin Sensitivity; Cardiovascular Risk Factor
MeSH Terms: conditions — Parasomnias; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Restriction (Experimental): Women will undergo 4 nights of sleep restriction treatment.
  Interventions: Behavioral: Sleep Restriction
- Habitual Sleep (Experimental): Women will undergo 4 nights of habitual sleep treatment.
  Interventions: Behavioral: Habitual Sleep

INTERVENTIONS:
Behavioral: Sleep Restriction — Women will be undergo 4 nights of sleep restriction.
  Arms: Sleep Restriction
Behavioral: Habitual Sleep — Women will be undergo 4 nights of habitual sleep.
  Arms: Habitual Sleep

SUMMARY:
Inadequate sleep is an independent risk factor for metabolic abnormalities (such as obesity, insulin resistance, and hyperglycemia). Women report sleep disruption during the menopause transition (perimenopause) and into the postmenopausal years. Sleep disruption is one of the primary reasons why midlife women seek medical care, with up to 60% reporting significant sleep disturbances (e.g., trouble falling asleep, early morning waking, and hot flashes/night sweats). Despite the majority of women experiencing sleep disruption, no study has investigated the molecular mechanisms linking sleep disruption and the changes in metabolism that coincide with menopause.

DETAILED DESCRIPTION:
The investigators will conduct a randomized, crossover trial investigating the effect of sleep restriction compared to habitual sleep on adipose tissue and skeletal muscle insulin sensitivity in vivo and ex vivo. The investigators will randomize up to 10 healthy postmenopausal women with overweight/obesity and ≥6.5 hours of self-reported habitual nightly sleep to 4 nights of each sleep condition (sleep restriction and habitual sleep). After the fourth night of each sleep condition, the investigators will administer a two-step hyperinsulinemic-euglycemic clamp and collect skeletal muscle and adipose tissue samples prior to insulin infusion.

The overarching hypothesis is that sleep restriction will reduce skeletal muscle and adipose tissue insulin sensitivity compared to habitual sleep.

ELIGIBILITY:
INCLUSION CRITERIA:

* Body mass index (BMI) 25-35 kg/m2 (inclusive)
* Postmenopausal (self-reported absence of menstrual cycle for 1-year)
* Within 10 years of final menstrual cycle
* Self-reported nocturnal time in bed of ≥6.5 hours per night (for ≥5 nights during a usual week)
* Willing to not take naps or engage in moderate-to-vigorous physical activity/exercise during both sleep conditions
* Willing to consume only the meals provided during both sleep conditions
* Willing to have adipose tissue and skeletal muscle biopsies
* Willing to have blood, as well as adipose and muscle tissue stored for future use

EXCLUSION CRITERIA:

* Unstable weight in the last 3 months [gain or loss ≥5% of body weight]
* History of clinically diagnosed diabetes or a fasting blood glucose >126 mg/dL
* History of polycystic ovary syndrome (PCOS)
* Currently taking antihypertension medication known to affect adipose tissue and skeletal muscle metabolism (e.g., diuretics may be allowed)
* Chronic use of systemic glucocorticoids
* Chronic use of atypical antipsychotic or bipolar medications
* Initiation of antidepressant medication within the last 3 months
* Previous bariatric surgery (or other surgeries) for obesity or weight loss
* Chronic use of prescription or 'effective' over-the-counter medications affecting sleep, circadian rhythms, or glucose metabolism †
* Chronic use of hormone replacement therapy
* History of clinically diagnosed sleep apnea
* Shift workers (e.g., individuals awake or working between Midnight and 5AM)
* Inability to spend 5 nights at Pennington Biomedical
* Unwilling to eat only the food and drink provided by study staff while in the study
* Unwilling to maintain a consistent and prescribed sleep schedule while in the study
* Unwilling to maintain a consistent eating schedule while in the study

Sporadic use of certain medications is fine (however, enrollment will depend on a case-by-case basis). If taking sporadically, women should not be taking the medication for 1-month prior to the first Run-In period.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Glucose infusion rate (via 2-step hyperinsulinemic-euglycemic clamp) (in vivo) | 4 days
  Insulin sensitivity by a 2-step hyperinsulinemic euglycemic clamp is performed at the end sleep conditions.

SECONDARY OUTCOMES:
Adipose tissue insulin sensitivity (via free fatty acid area-under-the-curve during the low-dose clamp) (in vivo) | 4 days
  During the low-dose insulin portion of the hyperinsulinemic-euglycemic clamp, free fatty acids will be samples across a 3-hour period to quantify a surrogate measure of adipose tissue insulin sensitivity in vivo.
Insulin-dependent suppression of lipolysis (via ex vivo adipose tissue biopsy analyses) | 4 days
  Release of free fatty acids and glycerol in culture.
Fat oxidation and substrate switching (via ex vivo skeletal muscle biopsy analyses) | 4 days
  Using primary myotubes, fat oxidation and substrate switching will be tested by measuring [1-14C]palmitate oxidation ± varying levels of glucose and pyruvate
Insulin sensitivity (via ex vivo skeletal muscle biopsy analyses) | 4 days
  Myotubes will be incubated ± insulin (100nM) in media containing: [U-14C]-glucose to measure glucose oxidation and glycogen synthesis; [3H]-2-deoxyglucose to assess glucose uptake; or unlabeled DMEM to test insulin signaling (western blot)
Gene expression (via ex vivo skeletal muscle biopsy analyses with RNASeq and RT-PCR) | 4 days
  Genes related to oxphos and circadian clock regulators will be assessed by RNASeq and confirmed with RT-PCR.
Glucose Area-Under-The-Curve (via 2-hour standard meal test) | 4 days
  Glucose area-under-the-curve (AUC) will be calculated throughout a 2-hour period following consumption of a standard meal (dinner shake) test on Day 4 of each sleep condition.
Insulin Area-Under-The-Curve (via 2-hour standard meal test) | 4 days
  Insulin area-under-the-curve (AUC) will be calculated throughout a 2-hour period following consumption of a standard meal (dinner shake) test on Day 4 of each sleep condition.
Blood pressure (via 24-hour ambulatory blood pressure monitoring) | 24 hours
  Blood pressure monitoring will be performed for a 24-hour period during Day 3 of each sleep conditions.
Resting metabolic rate (via indirect calorimetry) | 4 days
  O2 consumption and CO2 production will be measured by indirect calorimetry for 40 min (last 30 min will be used for calculations) using a metabolic cart. Resting metabolic rate will be derived using standard equations.

CONTACTS AND LOCATIONS:
Overall Officials: Kara L Marlatt, PhD, MPH, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Singh P, Beyl RA, Stephens JM, Noland RC, Richard AJ, Boudreau A, Hebert RC, Ravussin E, Broussard JL, St-Onge MP, Marlatt KL. Effect of sleep restriction on insulin sensitivity and energy metabolism in postmenopausal women: A randomized crossover trial. Obesity (Silver Spring). 2023 May;31(5):1204-1215. doi: 10.1002/oby.23739. Epub 2023 Mar 30. PMID 36998155